CLINICAL TRIAL: NCT00016796
Title: Language Stimuli Screening in Children
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010181; 01-N-0181
Record Dates: First submitted 2001-06-02; First posted 2001-06-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: Language Disorder; Healthy
Keywords: Reading; Naming
MeSH Terms: conditions — Language Disorders

SUMMARY:
This study will determine baseline language skills in children 4 to 8 years old. The data will be used to design studies using functional magnetic resonance imaging (fMRI) to identify what areas of the brain in children are involved in understanding language. This information is important for children who require brain surgery to control seizures.

Healthy normal volunteers between the ages of 4 and 8 years who have an IQ of 70 or more; who have no history of neurologic, psychiatric or language disorder; who are performing at or above grade level, and who are native English speakers may be eligible for this study.

Participants will be asked to do the following:

* name pictures or read words that appear on a computer screen
* listen to stories and answer questions about them
* match pictures to a spoken word

The children's responses will be recorded.

DETAILED DESCRIPTION:
We propose to study normal children to establish baseline data to use to develop novel sets of stimuli for functional imaging paradigms. Tasks using these stimuli will include object naming, sentence comprehension, and single word reading.

ELIGIBILITY:
INCLUSION CRITERIA:

Children will be between the ages 4 and 8 are eligible.

EXCLUSION CRITERIA:

Children who meet one of the following criteria are not eligible:

IQ below 70;

History of neurologic or psychiatric disorders;

History of an language disorder;

Performing below grade-level;

Non-native English speaker.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2001-05; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hertz-Pannier L, Gaillard WD, Mott SH, Cuenod CA, Bookheimer SY, Weinstein S, Conry J, Papero PH, Schiff SJ, Le Bihan D, Theodore WH. Noninvasive assessment of language dominance in children and adolescents with functional MRI: a preliminary study. Neurology. 1997 Apr;48(4):1003-12. doi: 10.1212/wnl.48.4.1003. PMID 9109891
- [Background] Devinsky O, Perrine K, Llinas R, Luciano DJ, Dogali M. Anterior temporal language areas in patients with early onset of temporal lobe epilepsy. Ann Neurol. 1993 Nov;34(5):727-32. doi: 10.1002/ana.410340517. PMID 8239568
- [Background] Cycowicz YM, Friedman D, Rothstein M, Snodgrass JG. Picture naming by young children: norms for name agreement, familiarity, and visual complexity. J Exp Child Psychol. 1997 May;65(2):171-237. doi: 10.1006/jecp.1996.2356. PMID 9169209